CLINICAL TRIAL: NCT03828409
Title: Comparison Of Post-operative Pain In Short Versus Long Stitch Technique For Abdominal Wall Closure After Elective Laparotomy- A Double-Blind, Randomized Controlled Trial
Brief Title: Comparison of Post-operative Pain in Short Versus Long Stitch for Laparotomy Closure
Acronym: Shortstitch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NMRR-16-1892-32723
Record Dates: First submitted 2019-01-28; First posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Pain, Postoperative
Keywords: short stitch; post-operative pain; PCA morphine usage; elective midline laparotomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two arms (short stitch: SS and long stitch:LS).The LS belongs to our conventional mass closure technique for midline laparotomy. SS technique has been used to investigate other parameters such as surgical site infection and incisional hernia.
  This study is carried out to evaluate if SS technique will reduce post-operative pain.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient will not know what technique was used for the abdominal wall closure. The medical officers that will assess patient's PCA morphine usage and VAS score post-operatively will not know which technique of suturing was used for that particular patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short stitch (Active Comparator): short stitch used as one arm
  Interventions: Procedure: Short stitch; Procedure: Long stitch
- Long stitch (Active Comparator): Long stitch as conventional mass-closure technique
  Interventions: Procedure: Short stitch; Procedure: Long stitch

INTERVENTIONS:
Procedure: Short stitch — The rectus sheath are cleaned off the subcutaneous fats. Short stitch technique uses smaller needle and suture material. The suture is placed nearer to each other as compared to our conventional long stitch technique. It has inter-suture distance of 5mm and 5mm distance from rectus edge. The suture will be started at one end and sutured continuous until the other end. Hence, this technique is applied without tension.
Procedure: Long stitch — Long stitch uses a larger needle and suture material. The suture is placed 1cm from the linea alba and 1 cm from previous suture. This technique include mass closure sutures at the midline laparotomy

SUMMARY:
Laparotomy is a surgical procedure where an incision is made through the abdominal wall in order to gain access to the peritoneal cavity. Midline laparotomy incisions were the main type of abdominal access. However, there were complications associated with laparotomy such as incisional hernia, post-operative pain, surgical site infection and burst abdomen. The anterior abdominal wall consists of skin, fascia, subcutaneous fat, external oblique aponeurosis, internal oblique muscles, transversus abdominis and rectus muscles. The skin and parietal peritoneum are supplied by T7- T12 and L1 nerve. Hence, breaching of the peritoneum, giving rise to post-operative laparotomy pain. It is reported that approximately 60% of patients who underwent laparotomy do complain of post-operative pain.

Techniques of abdominal wall closure has been constantly in order to develop an ideal suture technique to minimise wound complications. One of the most significant changes in abdominal closure technique was the introduction of mass closure technique, known as 'long stitch' (LS). This conventional mass closure, uses a suture-to-wound length ratio (SL:WL) of 4:1, achieved by the use of continuous sutures at one centimetre from rectus edge with inter-suture distance of one centimetre. Studies have shown LS caused compression of tissues enclosed in the mass stitch, leading to tissue ischaemia and necrosis. 'Short stitch' (SS) was introduced in 1980s where it was reported to result in lower rate of incisional hernia and surgical site infection. It has a SL:WL of more than four, achieved by placing the suture five millimetres from rectus edge with inter-suture distance of five millimetre as well. It incorporates only the linea alba, which may reduce tension and post-operative pain.Studies has indicate that approximately 40% of post-operative patients reported inadequate pain relief despite therapeutic intervention. Inadequate pain control is associated with complications such as atelectasis, prolonged immobilization and hospital stay, thromboembolic event, cardiac morbidity, insomnia, ileus and poor wound healing The Visual Analog Scale (VAS) of pain is commonly used as measures of pain score or intensity in clinical trials. A more objective way to evaluate the post-operative pain is to assess the usage of patient-controlled analgesia (PCA) over a period of time. The commonly used PCA drug for post-operative patient is morphine. As SS relies on less tension and proper distribution of force along the fascial plane, it is possible that it might reduce post-operative pain as compared to LS technique. It can be assessed using total usage of analgesia (intravenous infusion or PCA), with correlation to the respective visual-analogue scales (VAS) or numeric rating scales (NRS) at that particular time. There is no study that evaluate post-operative pain difference between SS and LS technique.

The hypothesis of this study is that SS will reduce PCA morphine usage after midline laparotomy, which translate into reduction in post-operative pain. In order to detect the 30% reduction of PCA morphine, 86 patients are required.

DETAILED DESCRIPTION:
Laparotomy is a surgical procedure where an incision is made through the abdominal wall in order to gain access to the peritoneal cavity. Midline laparotomy incisions were the main type of abdominal access However, there were complications associated with laparotomy such as incisional hernia, post-operative pain, surgical site infection and burst abdomen. The anterior abdominal wall consists of skin, fascia, subcutaneous fat, external oblique aponeurosis, internal oblique muscles, transversus abdominis and rectus muscles. The rectus abdominis muscles is covered by rectus sheath, formed by aponeurosis of the internal oblique muscles except posterior layer from the arcuate line downwards. The sheath contains the ends of the lower six thoracic nerves (T7-T12) with first lumbar nerve The skin and parietal peritoneum are supplied by T7- T12 and L1 nerve. Hence, breaching of the peritoneum, giving rise to post-operative laparotomy pain. It is reported that approximately 60% of patients who underwent laparotomy do complain of post-operative pain.

Techniques of abdominal wall closure has been constantly revised in order to develop an ideal suture technique to minimise wound complications. One of the most significant changes in abdominal closure technique was the introduction of mass closure technique, known as 'long stitch' (LS). This conventional mass closure, uses a suture-to-wound length ratio (SL:WL) of 4:1, achieved by the use of continuous sutures at one centimetre from rectus edge with inter-suture distance of one centimetre. Studies have shown LS caused compression of tissues enclosed in the mass stitch, leading to tissue ischaemia and necrosis. 'Short stitch' (SS) was introduced in 1980s where it was reported to result in lower rate of incisional hernia and surgical site infection. It has a SL:WL of more than four, achieved by placing the suture five millimetres from rectus edge with inter-suture distance of five millimetre as well. It incorporates only the linea alba, which may reduce tension and post-operative pain.

Effective post-operative pain management is an important aspect in surgical patient care. Studies has indicate that approximately 40% of post-operative patients reported inadequate pain relief despite therapeutic intervention. Inadequate pain control is associated with complications such as atelectasis, prolonged immobilization and hospital stay, thromboembolic event, cardiac morbidity, insomnia, ileus and poor wound healing. The Visual Analog Scale (VAS) of pain is commonly used as measures of pain score or intensity in clinical trials. A more objective way to evaluate the post-operative pain is to assess the usage of patient-controlled analgesia (PCA) over a period of time. The commonly used PCA drug for post-operative patient is morphine. As SS relies on less tension and proper distribution of force along the fascial plane, it is possible that it might reduce post-operative pain as compared to LS technique. It can be assessed using total usage of analgesia (intravenous infusion or PCA), with correlation to the respective visual-analogue scales (VAS) or numeric rating scales (NRS) at that particular time. There is no study that evaluate post-operative pain difference between SS and LS technique.

This is a prospective, multi-centered, double-blind randomized controlled trial to look into comparison of post-operative pain after elective laparotomy: short versus long stitch technique of closure in two tertiary hospitals. The study started in January 2017 and completed in November 2018. Patient who fulfilled the criteria of recruitment were included into this study.

In order to detect difference of 30% of PCA morphine usage, 86 patients are required. Both group of patients will received equal pre-operative analgesia, antibiotics and induction again. Patients will be randomized into LS and SS group. Once the aim of the surgery is achieved, the operating surgeon will open the sealed enveloped, which contain the group and technique of suture used. Postoperatively patient will be receiving oral paracetamol and taught on PCA morphine usage. PCA morphine usage and VAS score will be assessed by medical officer that are blinded to the treatment. Primary outcome is PCA morphine usage 24 hours post-surgery. Secondary outcome are presence of surgical site infection and length of hospital stay. Patients will subsequently be discharged by the surgeon in charge based on the discharge criteria. Patients will be follow-up in outpatient clinic on same interval. Presence of adverse events or complications will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Elective primary midline laparotomy,
* ASA Class I to III
* hemodynamically stable
* able to provide consent for surgery

Exclusion Criteria:

* Emergency laparotomy
* pregnancy
* history of previous midline laparotomy
* allergic to opiates
* unable to use PCA morphine (handicapped)
* patient will be planned for stoma creation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Reduction of PCA morphine usage post-operatively | 24 hours
  Measure total usage of PCA morphine

SECONDARY OUTCOMES:
Presence of Surgical site infection | throughout hospital stay, 2 weeks, 6 weeks and then 8 weeks during follow up (up to 1 year)
  Any surgical site infection at surgical site
Length of hospital stay | since day 1 hospital admission until the time when patient is deemed fit to be discharged (up to 1 month)
  number of days patient was admitted in the ward